CLINICAL TRIAL: NCT05278182
Title: A Placebo Controlled, Double-blind, Randomised Trial for Assessment of the Efficacy of Naoxintong Capsules in the Treatment of Coronary Atherosclerotic Plaque in Patients With Acute Myocardial Infarct on the Basis of Optimal Medical Therapy (Aspirin,Statins, Clopidogrel, Etc.)
Brief Title: A Study for Exploring the Efficacy of Naoxintong Capsules in the Treatment of Coronary Atherosclerotic Plaque on the Basis of Optimal Medical Therapy (Aspirin,Statins,Clopidogrel, Etc.): Stage One
Acronym: NXT-ASSESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Runlin Gao, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRFH20180010
Record Dates: First submitted 2022-02-06; First posted 2022-03-14 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: on the Basis of Optimal Medical Therapy
MeSH Terms: conditions — Atherosclerosis | interventions — naoxintong

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naoxintong Capsule (Experimental): Naoxintong Capsule
  Interventions: Drug: Naoxintong Capsule
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naoxintong Capsule — Patients with acute myocardial infarct on the basis of optimal medical therapy will take Naoxintong capsules following directions for 12 months
  Arms: Naoxintong Capsule
Drug: Placebo — Patients with acute myocardial infarct on the basis of optimal medical therapy will take placebo following directions for 12 months
  Arms: Placebo

SUMMARY:
To evaluate and compare the change of plaque composition by VH-IVUS imaging in subjects who take NXT and placebo in post-PCI of AMI patients during 12 months follow-up.

DETAILED DESCRIPTION:
NXT-ASSESS is a placebo controlled,double-blind,randomised trial for assessment of the efficacy of Naoxingtong capsules in the treatment of coronary atherosclerotic plaque in patients with acute myocardial infarct on the basis of optimal medical therapy.A total of approximately 80 AMI patients with selective PCI indication who take NXT and placebo in post-PCI 12 months

ELIGIBILITY:
Inclusion Criteria:

1. Signing informed consent;
2. Male or female aged 18 to 75 years old;
3. AMI patients with selective PCI indication primary PCI patients are exclusive;
4. No history of CABG or PCI;

Image inclusion criteria:

1. CCTA at least one in-segment ≥20% and ≤70% diameter stenosis non-culprit vessel in the proximal-middle segments of RCA, LCX, LAD (the proximal and distal plaque within 5mm, same as below);
2. Radiography diameter of target vessel, 2.5-4.0mm;
3. Studied vessel can be evaluated with OCT and IVUS; OCT: the visual target study lesion is lipid-rich plaque with lipid arc≥100 degree and fiber cap thickness≤120µm.

Exclusion Criteria:

1. Life expectancy is less than 1 year;
2. Cannot implant drug stent;
3. Received ≥4weeks systematic treatment of statin and other lipid-lowering drug in the 3 months before admission;
4. Received ≥4 weeks systematic treatment of any traditional Chinese medicine;
5. Known to have adverse reaction to ingredients of NXT capsule;
6. Patients with severe heart disease that CABG or selective PCI, heart transplantationSAVR/TAVR are required during the study(12 months);
7. LVEF<40%;
8. Drug uncontrollable recurrent and highly symptomatic arrhythmia such as ventricular tachycaidia, atrial fibrillation with rapid ventricular rate and paroxysmal supraventricular tachycardia in the 3 months before ACS admission;
9. Known any stroke;
10. Other operations arranged during the study period (12 months);
11. Uncontrollable hypertension, defined as resting systolic BP≥180mmHg;
12. Clinical confirmed as statin intolerance;
13. Type I diabetes or type 2 diabetes that is not well controlled;
14. Moderate and severe renal dysfunction (defined as eGFR<30ml/min/1.73m2);
15. Clinical confirmed liver disease or liver dysfunction (AST or ALT >3*ULN);
16. Clinical confirmed infection and other hematological, metabolic gastrointestinal or endocrine dysfunction that researchers believe not suitable for enrollment;
17. Known factors that may not be compliant, such as alcoholism, drug addiction, mental illness, etc.;
18. Participated in other clinical research projects, or within 30 days of the last participating clinical project;
19. Pregnant,breast feeding women or those plan to conceive during the study;
20. History of malignant tumor.

Lesion related:

1. Target segment severe calcification;
2. Failed PCI in culprit vessel;
3. Failed OCT screening (lipid arc/ fiber cap thickness does not match filter criteria);
4. Complications during the evaluation of OCT and IVUS/VH-IVUSOCT and IVUS/VH-IVUS evaluation failed due to instruments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Plaque composition | 12 months
  The change of plaque composition by virtual histology intravascular ultrasound imaging in subjects who take Naoxintong capsules and placebo in post-percutaneous coronary intervention follow-up
Plaque fibrous cap thickness | 12 months
  The change of plaque fibrous cap thickness measured by optical coherence tomography in subjects who take Naoxintong capsules and placebo during post-percutaneous coronary intervention follow-up

SECONDARY OUTCOMES:
Lipid arc | 12 months
  The change of lipid arc measured by optical coherence tomography in subjects who take Naoxintong capsules and placebo in post-percutaneous coronary intervention follow-up
Percent atheroma volume | 12 months
  The change of percent atheroma volume measured by intravascular ultrasound imaging in subjects who take Naoxintong capsules and placebo capsules during post-percutaneous coronary intervention follow-up
Total atheroma volume and low attenuation plaque volume | 12 months
  Total atheroma volume and low attenuation plaque volume measured by Coronary-CTA in subjects who take Naoxintong and placebo capsules during post-percutaneous coronary intervention follow-up
Lipid | 12 months
  The change of lipid measured by optical coherence tomography in subjects who take Naoxintong capsules
Platelet function | 12 months
  The change of platelet function measured by optical coherence tomography in subjects who take Naoxintong capsules
Clinical incidents | 12 months
  The number of clinical incidents in subjects who take Naoxintong capsules
Culprit vessel | 12 months
  The change of subjects culprit vessel with optical coherence tomography;

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing, Beijing Municipality, China